CLINICAL TRIAL: NCT04676282
Title: Psychological and Clinical Factors That Predict Intent to Deprescribe Medications Among Older Adults
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Maastricht University (Other); University of Iowa (Other); Johns Hopkins University (Other); Newcastle University (Other); University of Sydney (Other)
Responsible Party: Principal Investigator, Vordenberg, Clinical Associate Professor, University of Michigan
Other Study IDs: HUM00183129
Record Dates: First submitted 2020-12-09; First posted 2020-12-21 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Polypharmacy; Aging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (12):
- Survey 1 Statin - May cause harm: Participants in this arm will be exposed to a scenario in which a patient takes a statin (cholesterol) medication. The primary care provider raises the idea of stopping the statin as it may be causing harm.
  Interventions: Other: Hypothetical Scenario
- Survey 1 Stain - May lack benefit: Participants in this arm will be exposed to a scenario in which a patient takes a statin (cholesterol) medication. The primary care provider raises the idea of stopping the statin as it may lack benefit.
  Interventions: Other: Hypothetical Scenario
- Survey 1 Statin - May cause harm and lack benefit: Participants in this arm will be exposed to a scenario in which a patient takes a statin (cholesterol) medication. The primary care provider raises the idea of stopping the statin as it may be causing harm and lack benefit.
  Interventions: Other: Hypothetical Scenario
- Survey 1 PPI - May cause harm: Participants in this arm will be exposed to a scenario in which a patient takes a proton pump inhibitor (heartburn) medication. The primary care provider raises the idea of stopping the PPI as it may be causing harm.
  Interventions: Other: Hypothetical Scenario
- Survey 1 PPI - May lack benefit: Participants in this arm will be exposed to a scenario in which a patient takes a proton pump inhibitor (heartburn) medication. The primary care provider raises the idea of stopping the PPI as it may lack benefit.
  Interventions: Other: Hypothetical Scenario
- Survey 1 PPI - May cause harm and lack benefit: Participants in this arm will be exposed to a scenario in which a patient takes a proton pump inhibitor (heartburn) medication. The primary care provider raises the idea of stopping the PPI as it may be causing harm and lack benefit.
  Interventions: Other: Hypothetical Scenario
- Survey 2 Statin - May cause harm and lack benefit: Participants in this arm will be exposed to a scenario in which a patient takes a statin (cholesterol) medication. The primary care provider raises the idea of stopping the statin as it may be causing harm and lack benefit.
  Interventions: Other: Hypothetical Scenario
- Survey 2 Statin - Cardiologist: Participants in this arm will be exposed to a scenario in which a patient takes a statin (cholesterol) medication. The primary care provider raises the idea of stopping the statin previously started by a cardiologist.
  Interventions: Other: Hypothetical Scenario
- Survey 2 Statin - Daughter Preference: Participants in this arm will be exposed to a scenario in which a patient takes a statin (cholesterol) medication. The primary care provider raises the idea of stopping the statin but the patient's adult daughter prefers for her to continue the medication.
  Interventions: Other: Hypothetical Scenario
- Survey 2 Statin - Husband Stroke: Participants in this arm will be exposed to a scenario in which a patient takes a statin (cholesterol) medication. The primary care provider raises the idea of stopping the statin but the patient's husband previously had a stroke after he stopped his statin.
  Interventions: Other: Hypothetical Scenario
- Survey 2 Statin - Flier: Participants in this arm will be exposed to a scenario in which a patient takes a statin (cholesterol) medication. The primary care provider raises the idea of stopping the statin but the patient saw an educational flier about strokes in the waiting room.
  Interventions: Other: Hypothetical Scenario
- Survey 2 Statin - Difficulty Maintaining Lifestyle Changes: Participants in this arm will be exposed to a scenario in which a patient takes a statin (cholesterol) medication. The primary care provider raises the idea of stopping the statin but the patient recognizes that they have had difficulty exercising and eating healthier foods.
  Interventions: Other: Hypothetical Scenario

INTERVENTIONS:
Other: Hypothetical Scenario — Participants will be randomized to one of the arms. Each arm will contain a different hypothetical scenario.

SUMMARY:
The investigators are conducting two experimental surveys to explore clinical and psychological factors that influence older adults' willingness to stop medications in the face of polypharmacy.

DETAILED DESCRIPTION:
Around one-half of older adults take one or more medications that are inappropriate or medically unnecessary. These medications can cause side effects that are unacceptable to patients. Several studies provide guidance to clinicians about the process of stopping specific types of medications (e.g., steps that clinicians can take to reduce and stop a medication for anxiety or difficulty sleeping). However, these approaches are not always successful. A critical gap with these approaches is they tend to focus on the medication, rather than the patient, and their individual needs.

Our research team seeks to learn more about factors that are important to patients when they consider reducing or stopping a medication. The investigators will do this by conducting two surveys each with 4,800 older adults across four countries (United States, United Kingdom, Netherlands, and Australia). Each participant will be asked to give their opinions on a hypothetical patient scenario that has been developed by our diverse team in partnership with our stakeholder organizations. In the first survey, the investigators will examine how the reason for using the medication (e.g. preventing a disease or treating symptoms of a disease) as well as the reason for a recommendation to stop the medication (e.g. lack of benefit vs. potential for harm) influence older adults' willingness to stop medications. In the second survey, the investigators will examine how different social and clinical factors and whether the participant is making a recommendation about oneself (as if they were the patient in the case) or on behalf of the patient in the case (e.g., if it was their friend) influence their willingness to stop medications. The investigators will work with Qualtrics, an international company that distributes surveys, to collect this data that does not include any identifying information.

The investigators anticipate that once the survey is designed and show that it is successful for studying patient perspectives about stopping medicines, it can then apply the same study approach to test the effect of other relevant factor that may influence the decision to stop or reduce a medication. The investigators anticipate that our research will significantly contribute to our understanding of how older adults make decisions about stopping medications. This information will be helpful to researchers and clinicians to ensure future services can be developed to best support patients to make decisions about stopping or reducing inappropriate or unnecessary medication.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and older
* Resides in a participating country

Exclusion Criteria:

* None

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Adults 65 years and older who reside in a participating country
Sampling Method: Non-Probability Sample
Enrollment: 10184 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Response to question statement "I think that Mrs. EF should follow her PCPs recommendation and stop taking simvastatin." | 1 year
  Level of agreement with the primary care provider's recommendation to stop the medication presented in the hypothetical scenario (1=strongly disagree, 6=strongly agree)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weir KR, Marshall VD, Vordenberg SE. Latent Class Analysis Identifies Four Distinct Patient Deprescribing Typologies Among Older Adults in Four Countries. Innov Aging. 2025 Jan 17;9(2):igaf002. doi: 10.1093/geroni/igaf002. eCollection 2025. PMID 40008009
- [Derived] Vordenberg SE, Weir KR, Jansen J, Todd A, Schoenborn N, Scherer AM. Harm and Medication-Type Impact Agreement with Hypothetical Deprescribing Recommendations: a Vignette-Based Experiment with Older Adults Across Four Countries. J Gen Intern Med. 2023 May;38(6):1439-1448. doi: 10.1007/s11606-022-07850-5. Epub 2022 Nov 14. PMID 36376636